CLINICAL TRIAL: NCT03110861
Title: A Prospective, Multicenter, Single Arm Study to Evaluate the Safety and Effectiveness of Implantation of 'Transcatheter Pulmonary Valve (TPV)' for the Treatment of Congenital Heart Disease With Pulmonary Valve Disease
Brief Title: Pulsta® Transcatheter Pulmonary Valve Korean Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taewoong Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPV-101
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Congenital Heart Defect; Pulmonary Valve; Insufficiency, Congenital; Pulmonary Valve Stenosis
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Valve Stenosis | interventions — Replantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulsta® Transcatheter Pulmonary Valve (Experimental): Pulsta® Transcatheter Pulmonary Valve (TaeWoong Medical Co., Ltd. Korea)
  Interventions: Device: Pulsta® Transcatheter Pulmonary Valve (TPV) Replacement

INTERVENTIONS:
Device: Pulsta® Transcatheter Pulmonary Valve (TPV) Replacement — Pulsta® Transcatheter Pulmonary Valve Replacement

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the TPV in patients with pulmonary valve dysfunction.

DETAILED DESCRIPTION:
The TPV is indicated for use in patients with previous undergone replacement of bioprosthetic valve or conduit due to either pulmonary valve atresia, stenosis, regurgitation or a combination of them and present with dysfunctional right ventricular ourflow tract (RVOT) requiring treatment for severe pulmonary regurgitation and/or RVOT conduit obstruction. Consecutive subject data should be collected at discharge, 1, 3, 6 month, and 1-5 years post TPV implantation.

ELIGIBILITY:
Inclusion Criteria:

* Body weight greater than or equal to 30 kilograms
* Pulmonary regurgitation ≥moderate pulmonary regurgitation (PR) (≥3+) or RVOT conduit obstruction with mean gradient >35mmHg by echocardiography
* pulmonary artery annulus or in situ conduit size of ≥16 and ≤26mm
* Patient willing to provide written informed consent and comply with follow-up requirements

Exclusion Criteria:

* Pre-existing mechanical heart valve in any position
* Obstruction of the central veins (pulmonic bioprosthesis delivery system to the heart)
* Coronary artery compression
* A known hypersensitivity to Aspirin or Heparin
* Immunosuppressive disease
* Active infectious disease (e.g. endocarditis, meningitis)
* Estimated survival less than 6 months
* Female of child-bearing potential who are unable to take adequate contraceptive precautions, are known to be pregnant, or are currently breastfeeding an infant.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Hemodynamic functional improvement at 6month | 6 months
  Hemodynamic functional improvement is defined as mean RVOT gradient ≤30 mmHg by continuous wave doppler, and a pulmonary regurgitant fraction <20% by cardiac magnetic resonance (MR).
Procedural / Device related serious adverse events at 6month | 6 months

SECONDARY OUTCOMES:
Procedural success | 5 days
  Procedural success is defined as the TPV implant within desired position, Right ventricle-Pulmonary artery (RV-PA) peak systolic pressure gradient <35mmHg by catheter, less mild pulmonary regurgitation by angiography, and freedom from explantation of the TPV at 24 hours post-implant.
Hemodynamic function | 5 years
  Hemodynamic function will be measured including peak RVOT pressure gradient, mean RVOT pressure gradient, RV-PA pressure gradient, RV pressure, cardiac output, cardiac index, RV end-diastolic volume by echocardiography, cardiac MR, or catheterization.
Severity of pulmonary regurgitation | 5 years
New York Heart Association (NYHA) functional classification | 5 years
Stent fracture | 5 years
  Stent fracture will be assessed by the investigator through radiography (X-ray, Fluoroscopy).
Catheter reintervention on TPV | 5 years
Reoperation | 5 years
Procedural / Device related serious adverse events | 5 years
Death (all cause / procedural / device-related) | 5 years
Other adverse events | 5 years
Pulmonary regurgitant fraction | 6 months
  Pulmonary regurgitant fraction will be measured by cardiac MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Gi Beom Kim, phD. MD., Study Chair — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Seoul National University Hospital, Seoul, Haehak-ro Jongno-gu
  - Sejong General Hospital, Bucheon-si, Hohyun-ro, Sosa-gu
  - Samsung Medical Center, Seoul, Ilwon-ro, Gangnam-gu
  - Asan Medical Center, Seoul, Olympic-ro, Songpa-gu
  - Severance Hospital, Seoul, Yonsei-ro, Seodaemun-gu

IPD SHARING:
Plan to Share IPD: No